CLINICAL TRIAL: NCT02206503
Title: A PHASE II, MULTI-CENTER, OPEN LABEL STUDY OF CYCLOPHOSPHAMIDE IN MULTIPLE MYELOMA PATIENTS WITH BIOCHEMICAL PROGRESSION DURING LENALIDOMIDE-DEXAMETHASONE TREATMENT FOR RELAPSED/REFRACTORY MULTIPLE MYELOMA
Brief Title: Cyclophosphamide With Biochemical Progression During Lenalidomide-Dexamethasone Treatment for Relapsed/Refractory Multiple Myeloma (MM)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione EMN Italy Onlus (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRd
Record Dates: First submitted 2014-02-06; First posted 2014-08-01 (Estimated); Last update posted 2018-08-02 (Actual); Status verified 2018-08

CONDITIONS: Multiple Myeloma
Keywords: LENALIDOMIDE; BIOCHEMICAL PROGRESSION; RELAPSED/REFRACTORY MM; WITHOUT CRAB
MeSH Terms: conditions — Multiple Myeloma; Recurrence | interventions — Cyclophosphamide; Lenalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cyclophosphamide; Lenalidomide; Dexamethasone (Experimental): MM Patients who experienced biochemical progression during Rd treatment without CRAB (signs of organ damage, multiple myeloma-related, as renal impairment and/or anemia and/or new bone lesions and/or hypercalcemia), will continue:
  * Lenalidomide orally at the dose of 25 mg/day for 21 days every 28 days.
  * Dexamethasone orally at the dose of 40 mg once a week.
  Adding:
  · Cyclophosphamide orally at the dose of 50 mg/day on days 1-21 every 28 days. CRd combination will be continued for 9-4week cycles. Patients will not receive any maintenance therapy.
  Interventions: Drug: Cyclophosphamide; Drug: Lenalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Cyclophosphamide — This protocol is a phase II multicenter, open label study designed to determine whether the addition of Cyclophosphamide to Rd (CRd) treatment significantly increases response rates and prolonged the outcome (PFS, OS) in patients who experienced a biochemical relapse, without CRAB under Rd treatment. The treatment period includes: administration of the combination CRd for 9 cycles. In order to assess the efficacy and safety of treatment, patients will attend the study center visits at least every 2 weeks. The response will be assessed after each cycle. During the LTFU period, after development of confirmed PD, all patients are to be followed for survival every 1-3 months via telephone or office visit.
Drug: Lenalidomide
Drug: Dexamethasone

SUMMARY:
This study evaluates the efficacy of the addiction of Cyclophosphamide to Revlimid-low dose dexamethasone (Rd) in relapsed/refractory Multiple Myeloma patients, who experienced a biochemical progression, without CRAB, during Rd treatment.

DETAILED DESCRIPTION:
This protocol is a phase II multicenter, open label study designed to determine whether the addiction of Cyclophosphamide to Rd (CRd) treatment significantly increases response rates and prolonged the outcome (PFS, OS) in patients who experienced a biochemical relapse, without CRAB under Rd treatment. Patients will be evaluated at scheduled visits in up to 3 study periods: pre-treatment, treatment and long-term follow-up (LTFU).

The pre-treatment period includes: screening visits, performed at study entry. After providing written informed consent to participate in the study, patients will be evaluated for study eligibility. The screening period includes the availability of inclusion criteria described above. Subjects who meet all the inclusion criteria will be enrolled.

The treatment period includes: administration of the combination CRd for 9 cycles. In order to assess the efficacy and safety of treatment, patients will attend the study center visits at least every 2 weeks. The response will be assessed after each cycle.

During the LTFU period, after development of confirmed progression disease (PD), all patients are to be followed for survival every 1-3 months via telephone or office visit.

ELIGIBILITY:
Inclusion Criteria:

* Patient with relapse/refractory multiple myeloma who experienced biochemical progression, without CRAB, during treatment with Rd. CRAB means the presence of organ damage, multiple myeloma related (renal impairment and/or anemia and/or new bone lesions and/or hypercalcemia). It is sufficient one of the previous signs for defining the presence of CRAB. Biochemical progression means: positivization of serum/urine immunofixation for patients who reached a complete remission with Rd treatment or at least 25% increment of monoclonal component in serum/urine for patients who reached at least a stable disease (SD).
* Patient exposed to previous therapy included Lenalidomide, Thalidomide, Bortezomib and/or autologous stem cell transplantation (ASCT) and in treatment with Rd.
* Patient is, in the investigator(s) opinion, willing and able to comply with the protocol requirements.
* Patient has given voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to their future medical care.
* Female patient is either post-menopausal or surgically sterilized or, if at childbearing potential, must: understand that the study medication could have an expected teratogenic risk.
* Agree to use, and be able to comply with, effective contraception without interruption, 4 weeks before starting study drug, throughout study drug therapy (including dose interruptions) and for 4 weeks after the end of study drug therapy, even if she has amenorrhea. This applies unless the subject commits to absolute and continued abstinence confirmed on a monthly basis. The following are effective methods of contraception*:

  * Implant**
  * Levonorgestrel-releasing intrauterine system (IUS)**
  * Medroxyprogesterone acetate depot
  * Tubal sterilisation
  * Sexual intercourse with a vasectomised male partner only; vasectomy must be confirmed by two negative semen analyses
  * Ovulation inhibitory progesterone-only pills (i.e., desogestrel)
* Combined oral contraceptive pills are not recommended. If a subject was using combined oral contraception, she must switch to one of the methods above. The increased risk of venous thromboembolism (VTE) continues for 4 to 6 weeks after stopping combined oral contraception.
* **prophylactic antibiotics should be considered at the time of insertion particularly in patients with neutropenia due to risk of infection.
* Agree to have a medically supervised pregnancy test with a minimum sensitivity of 25 mills International Units on milliliter (mIU/ml) not more than 3 days before the start of study medication once the subject has been on effective contraception for at least 4 weeks. This requirement also applies to women of childbearing potential who practice complete and continued abstinence.
* Agree to have a medically supervised pregnancy test every 4 weeks including 4 weeks after the end of study treatment, except in the case of confirmed tubal sterilization. These tests should be performed not more than 3 days before the start of next treatment. This requirement also applies to women of childbearing potential who practice complete and continued abstinence.
* † A female subject or a female partner of a male subject is considered to have childbearing potential unless she meets at least one of the following criteria: Age

  ≥50 years and naturally amenorrhoeic for ≥ 1 year (amenorrhoea following cancer therapy does not rule out childbearing potential), premature ovarian failure confirmed by a specialist gynaecologist, previous bilateral salpingooophorectomy or hysterectomy, xy genotype, Turner's syndrome or uterine agenesis.
* Male subjects must:

  * Agree to use condoms throughout study drug therapy, during any dose interruption and for one week after cessation of study therapy if their partner is of childbearing potential and has no contraception.
  * Agree not to donate semen during study drug therapy and for one week after end of study drug therapy.
* All subjects must:

  * Agree to abstain from donating blood while taking study drug therapy and for one week following discontinuation of study drug therapy.
  * Agree not to share study medication with another person and to return all unused study drug to the investigator.
* Patient who obtain at least a SD with Rd treatment and experienced a biochemical progression without CRAB, during the treatment itself.
* Patient has a Karnofsky performance status ≥ 60%.
* Patient has a life-expectancy > 6 months.
* Patients must have a adequate cardiac function.
* Patients must have adequate pulmonary function.
* Patient has the following laboratory values within 14 days before Baseline (day 1 of the Cyclophosphamide):

  * Platelet count ≥ 50 x 109/L or ≥ 25 109/L if bone marrow involvement is ≥ 50% of plasma cells in bone marrow biopsy.
  * Absolute neutrophil count (ANC) ≥ 1.0 x 109/L or ≥ 0,5 109/L x if bone marrow involvement is ≥ 50% of plasma cells in bone marrow biopsy.
  * Corrected serum calcium ≤ 14 mg/dL (3.5 mmol/L).
  * Aspartate transaminase (AST): ≤ 2.5 x the upper limit of normal (ULN).
  * Alanine transaminase (ALT): ≤ 2.5 x the ULN.
  * Total bilirubin: ≤ 1.5 x the ULN.
  * Calculated or measured creatinine clearance: ≥ 30 mL/minute.

Exclusion Criteria:

* Patients with newly diagnosed multiple myeloma.
* Patients who relapsed from multiple myeloma with signs of organ damage related to disease (CRAB).
* Any serious medical condition, including the presence of laboratory abnormalities, which places the subject at an unacceptable risk if he or she participates in this study or confounds the experimental ability to interpret data from the study.
* Pregnant or lactating females.
* Prior history of malignancies, other than multiple myeloma, unless the subject has been free of the disease for ≥ 3 years. Exceptions include the following: Basal cell carcinoma of the skin, squamous cell carcinoma of the skin, carcinoma in situ of the cervix, carcinoma in situ of the breast, incidental histological finding of prostate cancer (TNM stage of T1a or T1b).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2015-04 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Efficacy in terms of response and survival | 2 years
  To assess the efficacy (response rate according to International Myeloma Working Group (IMWG) definition, appendix 2) after the addiction of Cyclophosphamide to Revlimid-Dexamethasone (CRd) in Multiple Myeloma patients, who experienced a biochemical progression during Rd treatment, without myeloma-related organ damage, CRAB.

SECONDARY OUTCOMES:
Safety in terms of hematological and non-hematological adverse events | 2 years
  The following evaluations will be conducted to assess the safety:
  * Adverse events
  * Concomitant medication and supportive therapies
  * Electrocardiogram and Chest Radiograph.
  * Medical history, physical examination, neurotoxicity assessment
  * Vital signs, body weight, height, and body surface area
  * Clinical laboratory evaluations (hematology, chemistry)
  * Health outcomes assessment
The progression free survival (PFS) | 2 years
The overall survival (OS) | 2 years
Duration of time to progression (TTP) | 2 years
Time to next therapy (TNT) | 2 years
Identification of patient's subgroups according to specific prognostic factors | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Maria Teresa Petrucci, MD, Principal Investigator — Policlinico Umberto I
Locations (1):
- Policlinico Umberto I, Rome, Italy